CLINICAL TRIAL: NCT04358003
Title: Plasma Adsorption in Patients With Confirmed COVID-19 Infection
Brief Title: Plasma Adsorption in Patients With Confirmed COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marker Therapeutics AG (Industry)
Collaborators: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH-007/B
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Failure; ARDS
Keywords: SARS-CoV-2; COVID-19; Spectra Optia Apheresis System; D2000 Cartridge; Terumo BCT; Marker Therapeutics
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Plasma Adsorption Cartridge (Experimental): Subjects will receive one treatment per day with the D2000 Cartridge for use with the Spectra Optia® Apheresis System (Optia SPD Protocol) for up to 4 hours (treatment cycle) for up to seven (7) days.
  Interventions: Device: Marker Therapeutics D2000 Cartridge (D2000) for use with the Spectra Optia® Apheresis System (Optia SPD Protocol)

INTERVENTIONS:
Device: Marker Therapeutics D2000 Cartridge (D2000) for use with the Spectra Optia® Apheresis System (Optia SPD Protocol) — Subjects will receive one treatment per day with the D2000 Cartridge for up to 4 hours (treatment cycle) for up to seven (7) days. Treatment may extend beyond 7 days, up to 14 days total, if deemed necessary and useful by the principal investigator (PI). Additional cartridges may be used, if needed, to achieve the maximum daily treatment duration of 4 hours. Each day, before initiating the treatment cycle, pre-treatment chemistry and hematology, coagulation status, and disease severity scores (SOFA, APACHE II) will be collected. Then, immediately following the therapy on each treatment day, post-therapy measurements will also be collected.
  Study Exit. Subjects will be exited from the study after the Day 28 follow-up visit which will occur 28 days after Study Day 1. Subjects will be included in the study for a total of 28 days. Subjects may also choose to discontinue at any time or conclude participation at the discretion of the PI or the subject's treating physician.

SUMMARY:
To characterize the ability of the D2000 Cartridge in combination with the Optia SPD Protocol to reduce the morbidity and mortality associated with SARS-CoV-2 infection in patients admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admitted to ICU
* Diagnosis of SARS-CoV-2 with any one of the following conditions:

  1. Early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS); or
  2. Severe disease, defined as:

     1. dyspnea,
     2. respiratory frequency ≥ 30/min
     3. blood oxygen saturation ≤ 93%
     4. partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or
     5. lung infiltrates > 50% within 24 to 48 hours; or
  3. Life-threatening disease, defined as:

     1. respiratory failure,
     2. septic shock, and/or
     3. multiple organ dysfunction or failure.
* Patient fact sheet is provided to the subject.
* Subject or legal representative is able and willing to give informed consent. If authorized by the IRB, emergent plasma adsorption with the D2000 cartridge may be initiated prior to consent.

Exclusion Criteria:

* Treatment limitation or a do not attempt to resuscitate in place
* Pregnancy
* Significant or uncontrolled bleeding
* In the opinion of the investigator, any other condition that precludes plasma adsorption with the D2000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Day 28

SECONDARY OUTCOMES:
Change in Sequential Organ Failure Assessment [SOFA] scores | Day 28
  Scale of 0-24 with a higher number indicating a worse outcome

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - UNM Health Science Center, Albuquerque, New Mexico
  - Providence Portland Medical Center, Portland, Oregon
  - Reading Hospital, West Reading, Pennsylvania
  - UT Southwestern/Clements Hospital, Dallas, Texas
  - UTMB, Galveston, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia

REFERENCES:
- [Derived] Choi C, De Simone N, Webb CB, Lahsaei P, Yates SG, Raval JS, Harkins MS, Hillebrand DJ, Belli A, Schlapobersky NA, Ipe TS, Banez-Sese GC, Khangoora VS, Nathan SD, Demko TM, Young DC, Caron S, Sarode R. Plasma Adsorption with the MTx.100 Column in Critically Ill COVID-19 Patients: A Prospective Study and Propensity Score Analysis. J Intensive Care Med. 2025 Mar;40(3):314-319. doi: 10.1177/08850666241280031. Epub 2024 Sep 12. PMID 39267408